CLINICAL TRIAL: NCT04908787
Title: A Randomized, Double-blind, Phase III Study of BD0801 Injection Combined With Chemotherapy Versus Placebo Combined With Chemotherapy in Patients With Recurrent, Platinum-resistant Epithelial Ovarian, Fallopian Tube , or Primary Peritoneal Cancer.
Brief Title: A Phase III Study of BD0801 Combined With Chemotherapy in Recurrent, Platinum-resistant Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Xianxiang Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM-63-OC-301
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Topotecan; Doxorubicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BD0801+chemotherapy (Experimental): BD0801 is in combination with one of three chemotherapies: Paclitaxel, Topotecan or Doxorubicin liposomes.
  Interventions: Drug: BD0801; Drug: Paclitaxel; Drug: Topotecan; Drug: doxorubicin liposome
- Placebo+chemotherapy (Placebo Comparator): Placebo is in combination with one of three chemotherapies: Paclitaxel, Topotecan or Doxorubicin liposomes.
  Interventions: Drug: Paclitaxel; Drug: Placebo; Drug: Topotecan; Drug: doxorubicin liposome

INTERVENTIONS:
Drug: BD0801 — Subjects receive BD0801 , intravenously, d1, d15, q4w, Dosage form: injectable, Strength: 1.5 mg/kg
  Arms: BD0801+chemotherapy
Drug: Paclitaxel — Subjects receive Weekly Paclitaxel, intravenously, d1, d8, d15, d22, q4w, Dosage form: injectable, Strength: 80 mg/m2
Drug: Placebo — Subjects receive Placebo, intravenously, d1, d15, q4w, Dosage form: injectable, Strength: 1.5 mg/kg
  Arms: Placebo+chemotherapy
Drug: Topotecan — Subjects receive Topotecan, intravenously, d1, d8, d15, q4w, Dosage form: injectable, Strength: 4mg/m2
Drug: doxorubicin liposome — Subjects receive doxorubicin liposome, intravenously, d1, , q4w, Dosage form: injectable, Strength: 40mg/m2

SUMMARY:
The standard systemic treatment for ovarian cancer is platinum-based chemotherapy. However, majority of patients relapse and eventually progress to platinum resistance. In patients with platinum-resistant or refractory ovarian cancer, effective treatment options are limited and the prognosis is very poor. Angiogenesis is essential for tumor growth and metastasis, and VEGF/VEGF receptor(VEGFR) signaling pathway is the most promising angiogenic target. This study aim to assess the efficacy and safety of the combination BD0801 and chemotherapy in patients with platinum-resistant recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >/=18 years of age;
* epithelial ovarian, fallopian tube or primary peritoneal cancer;
* platinum-resistant disease (disease progression within <6 months of platinum therapy)
* Eastern Cooperative Oncology Group（ECOG）performance status of 0-1

Exclusion Criteria:

* non-epithelial tumours
* ovarian tumours with low malignant potential
* Received 1 line of systemic therapy for ovarian cancer following platinum resistance and/or > 1 line of non-platinum systemic therapy prior to platinum resistance.
* prior radiotherapy to the pelvis or abdomen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Progression free survival(PFS) by blinded independent review committee(BIRC) | 2 year
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the IRC according to the RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall Survival (OS) | 2.5 year
  OS is the time interval from the date of randomization to death from any cause.
PFS by investigator | 2 year
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the investigator according to the RECIST1.1 criteria
Objective Response Rate (ORR) by investigator | 2 year
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by investigator according to RECIST 1.1 criteria
Disease Control Rate (DCR) by investigator | 2 year
  Proportion of subjects who have a complete or partial response, or stable disease relative to baseline as assessed by investigator according to RECIST 1.1 criteria
Objective Response Rate (DOR) by investigator | 2 year
  Measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria.
ORR by BIRC | 2 year
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by BIRC according to RECIST 1.1 criteria
DCR by BIRC | 2 year
  Proportion of subjects who have a complete or partial response, or stable disease relative to baseline as assessed by BIRC according to RECIST 1.1 criteria
DOR by BIRC | 2 year
  Measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria.
The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 2.5 year
  Frequency and severity of Adverse Events or Serious Adverse Events as defined by CTCAE version 5.0
Quality Of Life (QoL) | 2.5 year
  use European Organisation for Research and Treatment of Cance（EORTC）- QLQ-C30 questionnaire
Quality Of Life (QoL) | 2.5 year
  use EORTC-QLQ-OV28 questionnaire
Serum drug concentrations of BD0801 | 2 year
  Serum drug concentrations of BD0801 will be calculated.
rate of immunogenicity positive reaction | 2 year
duration of immunogenicity positive reaction | 2 year

CONTACTS AND LOCATIONS:
Locations (55):
- China (55):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - The First Affiliated Hospital of USTC West District,Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Cancer Hospital Chinese Academy Of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Guangxi Medical University Cancer Hospital&Guangxi Cancer Institute, Guangxi Cancer Hospital&Medical University School&Cancer Center, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Affiliated Cancer Hospital of Zhengzhou University and Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nanjing Women and Children's Healthcare Hospital, Women's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nantong Cancer Hospital, Nantong, Jiangsu
  - Xuzhou Central Hospital(Southeast University Affiliated Hospital), Xuzhou, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Norman Bethune Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Fukuang General Hospital of Liaoning Health Industry Group, Fushun, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital & Institute, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Center Hospital of Gynecology Obstetrics, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No